CLINICAL TRIAL: NCT02033798
Title: Impact of Medical Treatment for Benign Prostatic Hyperplasia on Chronic Renal Failure
Brief Title: The Effect of Daily Tamsulosin 0.2mg Administration on Renal Function in Patients With Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Seung-Ju Lee, Senior researcher, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L201401N2
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Kidney Failure; Prostatic Hyperplasia
Keywords: Urodynamics; Glomerular Filtration Rate
MeSH Terms: conditions — Kidney Failure, Chronic; Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamsulosin (Experimental): The dosage form of Tamsulosin is tablet, dosage is 0.2mg, frequency is once daily and duration is 6 months.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — Once Daily 0.2mg per oral for 6 months
  Other Names: Harnal D; Tamsnal

SUMMARY:
The purpose of this study is to determine whether medical treatment for bladder outlet obstruction is effective in improvement of glomerular filtration rate and/or proteinuria.

DETAILED DESCRIPTION:
Urodynamic parameters including maximal flow rate, compliance (infused volume gradient divided by bladder pressure gradient during cystometry), maximal detrusor pressure, bladder outlet obstruction index and Schäfer grade will be checked.

Estimated glomerular filtration rate and urinary protein to creatinine ratio will be checked.

International prostate symptom score will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Men with low urinary tract symptoms aged between 40 and 80
* Estimated glomerular filtration rate < 60 or evidence of proteinuria
* Bladder outlet obstruction index > 40, Schäfer grade 2 or more, maximal flow rate lower than 10 cc/s or postvoid residual urine > 100cc

Exclusion Criteria:

* Bladder outlet obstruction index less than 40, Schäfer grade 0 or 1, maximal flow rate higher than 10 ml/s and postvoid residual urine less than 100cc
* Want surgical procedure
* Evidence of prostate cancer or bladder cancer
* Major depressive disorder, Dementia, Parkinson's disease or neurological deficits
* History of pelvic irradiation
* Uncontrolled diabetes mellitus or hypertension
* Symptomatic orthostatic hypotension

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Maximal flow rate | 6 months
  This parameter can be obtained from urodynamic study.
Maximal detrusor pressure | 6 months
  This parameter can be obtained from urodynamic study.
Bladder outlet obstruction index | 6 months
  This parameter can be obtained from urodynamic study.
schäfer grade | 6 months
  This parameter can be obtained from urodynamic study.
Compliance | 6 months
  This parameter can be obtained from urodynamic study.

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | 6 months
Urinary protein to creatinine ratio | 6 months

OTHER OUTCOMES:
International prostate symptom score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Ju Lee, MD, PhD, Study Chair — The Catholic University of Korea; Dong Sup Lee, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea